CLINICAL TRIAL: NCT00785109
Title: Vitamin K Containing Nutritional Supplement for Activation of Matrix-GIa-proteins (MGP) and Inhibition of Aortic Valve Calcification Process
Brief Title: Vitamin K Supplement for Inhibition of the Progress in Aortic Valve Calcification
Acronym: 08-002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin K Study; 2008-005306-39
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Aortic Valve Calcification
Keywords: aortic valve calcification; vitamin K supplementation
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 100 patients daily additional intake of 2mg vitamin k1
  Interventions: Dietary Supplement: Vitamin K supplementation
- 2 (Placebo Comparator): 100 patients no additional intake of vitamin K
  Interventions: Dietary Supplement: Vitamin K supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin K supplementation — Daily vitamin K supplementation per os (2 mg once a day)Experimental 1 Placebo Experimental 2

SUMMARY:
In this mono-center,open,three-armes, controlled, randomized phase I study the progress of aortic valve calcification with and without vitamin K supplementation will be investgated. This will be done by means of measurements of concentrations from osteocalcine and MPG in blood serum, echocardiography, cardiac computed tomography and cardiac MRI

DETAILED DESCRIPTION:
Patients will be allocated to two groups with either

1. additional intake of 2 mg vitamin k1 daily
2. controll group without additional intake of Vitamin K

Treatment group a will include 100 patients, the controll group should include 100 patients. None of all patients should require renal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve calcification,verified by echocardiography

Exclusion Criteria:

* chronic or acute intestinal diseases
* terminal renal failure
* allergic reaction on soya containing products
* recent additional intake of vitamin K
* oral anticoagulation with vitamin K antagonists (Marcoumar)
* systemic therapy with corticosteroids
* anamnestic venous thrombosis (pelvet or legs)or embolization of lung arteria
* pregnant or breastfeeding women
* persons without mental ability or capacity to understand and follow the instructions of the investigator
* women of childbearing age without safe contraceptional devices
* minority

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Decrease of aortic valve calcification by activation of the calcification inhibiting protein MGP by means of additional intake of vitamin K | 18 months

SECONDARY OUTCOMES:
progression of diastolic and systolic dysfunction in the three treatment groups | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Koos, MD, Principal Investigator — RWTH Aachen University Departement of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonology and Vascular Medicine, Aachen, North Rhine-Westphalia, Germany